CLINICAL TRIAL: NCT05223946
Title: Treatment and Companion Diagnostics of Lower Back Pain Using SCENAR and Passive Medical Radiometry (MWR)
Acronym: SCENAR/MWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyrgyz State Medical Academy (Other)
Collaborators: Rostov State Medical University (Unknown); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1/13 24.01.2013
Record Dates: First submitted 2021-08-17; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-12

CONDITIONS: Low Back Pain, Recurrent
Keywords: Lower Back Pain; passive medical radiometry (MWR); SCENAR
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Microwave Radiometry (Active Comparator): Diagnostic Test: Passive Microwave Radiometry The MWR2020 (former RTM-01-RES) device is a unique commercially available CE marked device. The device is already registered in Russia and Kyrgyzstan for diagnostics of different diseases.
  Interventions: Diagnostic Test: Microwave Radiometry; Combination Product: Traditional Combination Therapy
- SCENAR (Experimental): Percutaneous electroneurostimulation (TENS) using the Self Controlled Energy Neuro Adaptive Regulator SCENAR-CHENS-01 device (ZAO OKB RITM, Taganrog, Russia)
  Interventions: Diagnostic Test: Microwave Radiometry; Device: SCENAR-CHENS-01; Combination Product: Traditional Combination Therapy

INTERVENTIONS:
Diagnostic Test: Microwave Radiometry — The MWR 2020 (former RTM-01-RES) device is a unique commercially available CE marked device. The device is already registered in Russia and Kyrgyzstan for diagnostics of different diseases. There were several works on identification of excess of microwave emission due to inflammatory, process, cancer and other disorders.
  Other Names: MWR
Device: SCENAR-CHENS-01 — Percutaneous electroneurostimulation (TENS) using the Self Controlled Energy Neuro Adaptive Regulator SCENAR-CHENS-01 device (ZAO OKB RITM, Taganrog, Russia)
  Arms: SCENAR
Combination Product: Traditional Combination Therapy — ketoprofen, tolperisone, symptomatic slow-acting drugs in osteoarthritis - SYSADOA - (glucosamine + chondroitin sulfate )

SUMMARY:
Evaluation of the effectiveness of treatment of nonspecific pain in the lower back (LBP) is currently largely based on the patient's subjective feelings. The purpose of this study was to use passive medical radiometry (MWR) as a tool for assessing the effectiveness of various treatment methods in patients with acute and subacute nonspecific LBP. Patients with pain assessment on a visual analogue scale (VAS) from 6 to 10 points were divided into 2 groups: Group I included patients with pharmacological, syndrome-oriented treatment (n = 30, age 54.9 ± 2.3 years); Group II is a combination pharmacotherapy with self-controlled energy-neuro-adaptive regulation (SCENAR) (n = 25, age 52.8 ± 2.5 years). The investigators will compare that the addition of SCENAR therapy (Group II) will be able to potentiate the analgesic effect of the treatment using VAS. the investigators will confirm that the thermal asymmetry visualization allows to identify the area of pathological muscle spasm and/or inflammation in the projection of the vertebral-motor segment.

DETAILED DESCRIPTION:
According to the Global Burden of Disease Study (2015), low back pain (LBP) has been one of the five leading causes of disability over the past 30 years. Indirect costs of unfulfilled work and social benefits are several times higher than the costs of actual treatment. In the "internal" structure of the LBP, nonspecific or musculoskeletal pain accounts for up to 80-90% of cases. LBP is characterized by a significant prevalence, high material costs for rehabilitation, and a large polymorphism of clinical manifestations. The number of treatment and diagnostic methods with a well-founded evidence base was very small. The main assessment of the effectiveness of therapy in most cases is based on the patient's subjective feelings and data from various questionnaires and scales. Subjunctivization of therapy evaluation leads to the underestimation of many treatment methods, which are questioned from the standpoint of evidence-based medicine. With this type of back pain, during clinical examination, radiography and MRI are inappropriate because of the lack of correlation between the severity of degenerative changes in the spine and the clinical picture.

It is the presence of pain that causes people to suffer, reduces the quality of life, and therefore non-steroidal analgesic drugs remain the drugs of the "first level". However, participants simultaneously have, especially with uncontrolled use, side effects on the gastrointestinal tract, cardiovascular, genitourinary systems, and other organs and systems.

Non-drug therapy is an important curative factor. One of the positively proven additional methods of treatment for various pain syndromes is percutaneous (transcutaneous) electro neurostimulation (TENS). The Cochrane Review showed the efficacy of TENS for acute pain of various origins. A comparative analysis with placebo was given with recommendations to consider TENS as a method of treatment, prescribed alone or in combination with other therapies. The method was also effective in treating neck pain in patients with whiplash injury after car accidents.

In addition to the subjective methods of assessing various methods and diagnostics of LBP treatment, passive medical radiometry (MWR) was chosen. The method is based on measuring the intensity of its own electromagnetic radiation of the internal tissues of the body in the ultrahigh-frequency range. MWR is widely used worldwide for various pathological conditions. It is known that processes occurring in the tissues of the body, especially those associated with pain, are often accompanied by a universal pathophysiological reaction. One of the signs of inflammation is an increase in temperature, which is associated with metabolic, vascular, and/or regulatory processes. Stable temperature changes precede or accompany clinical and morphological manifestations of the pathological process. Therefore, with a high probability, MWR can be used for early diagnosis and objective monitoring of treatment effectiveness.

Goal To evaluate the effectiveness of SCENAR treatment and MWR of various therapeutic regimens in patients with acute and subacute nonspecific LBP.

Materials and methods

The study is being carried out at the "Problematic Scientific Laboratory of Physical Methods of Diagnosis and Treatment" of Rostov State Medical University. A clinical randomized, parallel, divided into two groups (group selection method, even or odd), controlled, prospective study of patients with LBP is carried out. The local independent ethical committee of Rostov State Medical University approved the study (protocol No. 10/19 of 05/30/2019), and informed consent was obtained from all patients.

The total duration of the disease in patients ranged from 2 to 20 years, and the current exacerbation ranged from 1 d to 3 months. Clinical and neurological examination of patients with LBP is performed according to a specially developed protocol. The protocol included personal data, anamnestic data (including the duration of the current exacerbation), concomitant diseases, objective data, neurological status (including possible symptoms of radiculopathy and myelopathy), and a questionnaire for diagnosing neuropathic pain (Douleur Neuropathique en 4 questions - DN4). The inclusion criteria included patients with acute and subacute LBP of the musculoskeletal, nociceptive (with the duration of the current exacerbation up to 3 months inclusive), nonspecific character, caused by various degenerative-dystrophic lesions of the spine or paravertebral tissues (without specifying the source of pain) who were in outpatient or inpatient departments. The exclusion criteria included the presence of radiculopathy and myelopathy, known congenital anomalies of the spine, ankylosing spondylitis, reactive arthritis, rheumatoid arthritis, suspicion of a secondary nature of pain, gross cardiac arrhythmias, and probable neuropathic pain. Before treatment, some patients undergo MRI of the spine without axial load to exclude other diseases of the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* acute and subacute LBP of the musculoskeletal,
* nociceptive (with the duration of the current exacerbation up to 3 months inclusive),
* nonspecific character, caused by various degenerative-dystrophic lesions of the spine or paravertebral tissues (without specifying the source of pain) who were in outpatient or inpatient departments

Exclusion Criteria:

* presence of radiculopathy and myelopathy,
* known congenital anomalies of the spine,
* ankylosing spondylitis,
* reactive arthritis,
* rheumatoid arthritis,
* suspicion of a secondary nature of pain,
* gross cardiac arrhythmias, and probable neuropathic pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score (VAS) for pain for participants with traditional pharmacotherapy with the Self Controlled Energy Neuro Adaptive Regulator SCENAR-CHENS-01 device and traditional pharmacotherapy only. | 30 days
  Visual Analog Score for pain for Participants with TRADITIONAL treatment only (ketoprofen, tolperisone, symptomatic slow-acting drugs in osteoarthritis - SYSADOA - (glucosamine + chondroitin sulfate ) and COMBINED treatment (TRADITIONAL + SCENAR-CHENS-01) assessed using Visual Analog Score for pain.
  The Visual Analog Scale (VAS) is most commonly a straight 100-mm line, without demarcation, that has the words "no pain" at the left-most end and "worst pain imaginable" (or something similar) at the right-most end. The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Goryanin, PhD, Study Chair — MMWR LTD
Locations (2):
- Kyrgyzstan (2):
  - Educational - clinical - scientific medical center of KSMA, Bishkek, Chui
  - Batyr Osmonov, Bishkek

REFERENCES:
- [Background] Lanas A, Boers M, Nuevo J. Gastrointestinal events in at-risk patients starting non-steroidal anti-inflammatory drugs (NSAIDs) for rheumatic diseases: the EVIDENCE study of European routine practice. Ann Rheum Dis. 2015 Apr;74(4):675-81. doi: 10.1136/annrheumdis-2013-204155. Epub 2013 Dec 18. PMID 24351518
- [Background] Johnson MI, Paley CA, Howe TE, Sluka KA. Transcutaneous electrical nerve stimulation for acute pain. Cochrane Database Syst Rev. 2015 Jun 15;2015(6):CD006142. doi: 10.1002/14651858.CD006142.pub3. PMID 26075732
- [Background] Goryanin I, Karbainov S, Shevelev O, Tarakanov A, Redpath K, Vesnin S, Ivanov Y. Passive microwave radiometry in biomedical studies. Drug Discov Today. 2020 Apr;25(4):757-763. doi: 10.1016/j.drudis.2020.01.016. Epub 2020 Jan 28. PMID 32004473
- [Result] Lee TH, Kim SJ, Lim SM. Prevalence of disc degeneration in asymptomatic korean subjects. Part 2 : cervical spine. J Korean Neurosurg Soc. 2013 Feb;53(2):89-95. doi: 10.3340/jkns.2013.53.2.89. Epub 2013 Feb 28. PMID 23560172